CLINICAL TRIAL: NCT03713697
Title: Self-Collection and HPV Testing in Unscreened Women: a Feasibility Study in Brazil
Brief Title: Self-Collection and Human Papillomavirus (HPV) Testing in Unscreened Women: a Feasibility Study in Brazil
Acronym: HPV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Isabel Scarinci, Primary Investigator, University of Alabama at Birmingham
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: X150303007; P30CA013148 (NIH)
Record Dates: First submitted 2018-10-18; First posted 2018-10-22 (Actual); Last update posted 2018-10-22 (Actual); Status verified 2018-10

CONDITIONS: Cervical Cancer
Keywords: self-collection for HPV testing
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Vaginal Smears

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pap testing (Experimental): Women assigned to this arm were invited to get a Pap testing at the Basic Health Unit
  Interventions: Behavioral: Pap testing
- Self-Collection for HPV testing (Experimental): Women assigned to this arm were provided with a kit to engage in self-collection for HPV testing
  Interventions: Behavioral: Self-collection for HPV testing
- Choice (Experimental): Women assigned to this arm were given a choice between a Pap testing at the local Basic Health Unit or self-collection for HPV testing
  Interventions: Behavioral: Choice

INTERVENTIONS:
Behavioral: Pap testing — Un/underscreened women received a home visit by a Community Health Worker and were scheduled an appointment for a Pap testing at the Basic Health Unit
  Arms: Pap testing
Behavioral: Self-collection for HPV testing — Un/underscreened women received a home visit by a Community Health Worker and were given a kit to self-collect their own sampling for HPV testing at home
  Arms: Self-Collection for HPV testing
Behavioral: Choice — Un/underscreened women received a home visit by a Community Health Worker and were given a choice between scheduling an appointment for a Pap testing at the Basic Health Unit or self-collect their own sampling for HPV testing at home
  Arms: Choice

SUMMARY:
Our long-term goal is to decrease cervical cancer incidence and mortality among women in low- and middle-income countries (LMICs) by using the most efficacious and acceptable screening method, particularly among women who do not come to the clinic for their regular Pap testing. The purpose of this feasibility study is to compare three cervical cancer screening modalities (self-collection and HPV testing, Pap testing at the public health clinic, and choice between self-collection and HPV testing and Pap testing) among women who have not undergone cervical cancer screening within the past four years using a theory-based, culturally relevant intervention implemented by Community Health Workers (CHWs) via door-to-door visits. Three Basic Health Units (BHUs) within the public health system will be randomly assigned to one of the three screening modalities/conditions (self-collection and HPV testing, Pap testing at the local public health clinic, and choice between self-collection and HPV testing and Pap testing). CHWs will invite women who report not having been screened for cervical cancer in the past four years to participate in the study, and deliver a brief educational/behavioral session on cervical cancer and screening using a door-to-door approach under of one of the three conditions. The primary outcome will be adherence to cervical cancer screening. We hypothesize that (1) Women in the "choice" and "self-collection" groups will be more likely to engage in cervical cancer screening and display higher satisfaction with their screening than women assigned to the "Pap" with women assigned to the "choice" group having the highest adherence of the three groups; and (2) Within the "choice" group, more women will choose and complete self-collection than Pap test.

ELIGIBILITY:
Inclusion Criteria:

* No personal history of cervical cancer
* Not have engaged in cervical cancer screening for the past 4 years

Exclusion Criteria:

* None

Ages: 25 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 484 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2016-11-30 (Actual); Study Completion 2017-01-20 (Actual)

PRIMARY OUTCOMES:
Adherence to cervical cancer screening | baseline to 30 days
  Adherence to cervical cancer screening by completing either the Pap testing or self-collection for HPV testing)

CONTACTS AND LOCATIONS:
Overall Officials: Isabel C Scarinci, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- Universidade Estadual de Maringá, Maringá, Paraná, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Castle PE, Silva VRS, Consolaro MEL, Kienen N, Bittencourt L, Pelloso SM, Partridge EE, Pierz A, Dartibale CB, Uchimura NS, Scarinci IC. Participation in Cervical Screening by Self-collection, Pap, or a Choice of Either in Brazil. Cancer Prev Res (Phila). 2019 Mar;12(3):159-170. doi: 10.1158/1940-6207.CAPR-18-0419. Epub 2019 Jan 16. PMID 30651294